CLINICAL TRIAL: NCT05877534
Title: Effects of Individual Tailored Physical Exercise in Patients With Post COVID-19 Condition, Diagnosed With Postural Orthostatic Tachycardia Syndrome (POTS) - a Randomized Controlled Study
Brief Title: Effects of Individual Tailored Physical Exercise in Patients With POTS After COVID-19 - a Randomized Controlled Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Nygren-Bonnier, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-POTS-ReCov
Record Dates: First submitted 2023-05-24; First posted 2023-05-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Postural Orthostatic Tachycardia Syndrome; COVID-19; Post COVID-19 Condition; Post-Acute COVID-19 Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A 16 week period of exercise, supervised by a physiotherapist once a week. The exercise should be individually tailored from a programme based on a previous feasibility study. The program consist of exercises both to improve endurance and muscle strength. Progression and adjustments of time and position will be performed during the intervention period based any symptoms the participant exhibits. Progression should be halted if the participant experience PEM or other symptoms within >24hours after last exercise. The participants will also recieve standard care during the intervention period. Standard care includes (but not restricted to) information about POTS and lifestyle changes that may effect the symptoms, advice about fluid intake and nutrition, compression garments, pharmacological interventions etc.
  Interventions: Other: Individual tailored exercise
- Control (No Intervention): Standard care during 16 weeks. Standard care includes (but not restricted to) information about POTS and lifestyle changes that may effect the symptoms, advice about fluid intake and nutrition, compression garments, pharmacological interventions etc.

INTERVENTIONS:
Other: Individual tailored exercise — A 16 week period of progressive exercise, supervised by a physiotherapist once a week.
  Arms: Intervention

SUMMARY:
Covid-19 has the potential to affect physical, cognitive and psychological functions in multiple ways. It has been clear that a significant proportion of patients with Covid-19 develop long-term symptoms. The term post COVID-19 condition (defined by WHO) is used to describe the wide range of prolonged symptoms following the infection. Patients may need specialized rehabilitation to be able to meet the complex symptoms and problems that may arise. A more specific syndrome that seems to occur more frequently than expected in the group of non-hospitalized patients with post COVID-19 condition is the postural orthostatic tachycardia syndrome (POTS).

A randomized controlled design will be used to evaluate the effects of individual tailored physical exercise in patients with POTS after Covid-19.

Participants: Adults (>18 years) with post COVID-19 condition and diagnosed with POTS (n=60) will be included. Exclusion criteria: known pregnancy, cancer, already ongoing individual physical exercise (specific for POTS), or not able to perform measurements and/or intervention.

Procedure and outcomes: The primary outcomes are objectively measured time in upright position and health-related quality of life. Secondary outcomes are: physical activity, physical capacity, work ability and disease specific symptoms measured with tests and questionnaires.

Prior to randomization baseline measurements will be performed, aswell as after 16 weeks, 6 months and 12 months.

Intervention: Participants randomized to intervention will receive standard care and undergo a individually designed physical exercise program during 16 weeks, supervised and guided by a physiotherapist. The intervention will consist of different exercises to enhance muscle strength and endurance. Progression will be according to a program (based on previous feasibility studie) but should be halted if post exertional malaise (PEM) or other problems occur.

Controls: Participants randomized to control will receive standard care during 16 weeks.

Measurements of both groups (control and intervention) will be repeated after completion of a period of 16 weeks.

DETAILED DESCRIPTION:
Introduction:

Covid-19, was in March 2020, declared a global pandemic by the World Health Organization (WHO). In August 2021, in Sweden, over 1 100 000 cases were confirmed and over 14 000 deaths. Initially, it was suspected that Covid-19 would primarily affect the airways, but several studies have now shown that it is a disease with multisystem manifestations. The impact of the virus ranges from an asymptomatic infection to a severe and life-threatening disease that can affect the cardiac, renal gastrointestinal, nervous, endocrine, and musculoskeletal systems. Therefore, Covid-19 has the potential to affect physical, cognitive, and psychological functions in multiple ways.

It has been clear that a significant proportion of patients with Covid-19 develop long-term symptoms. Signs and symptoms may arise from any system in the body, often with significant overlap, and may develop over time. The term post COVID-19 condition (defined by WHO) is now used to describe the wide range of prolonged symptoms following the infection. Fatigue, decreased physical and psychological function have been reported in the initial recovery phase, but still little is known on the long-term consequences. Previous studies on the recovery and rehabilitation after other coronavirus shows the importance to develop tailored interventions.

A more specific syndrome that seems to occur more frequently in non-hospitalized persons with post COVID-19 condition is the postural orthostatic tachycardia syndrome (POTS). It is a chronic orthostatic intolerance where upright posture is associated with an excessive increase in heart rate (HR) and associated symptoms, such as palpitation, exercise intolerance, hypermobile joints, migraine headaches, brain-fog, sleep disturbances, and fatigue. Symptoms can be exacerbated by simple activities of daily life and the patients often report a low quality of life, equivalent to what patients with severe heart failure or COPD report. Consequently, patients seem to reduce their physical activity, which make them deconditioned and limits the activities in daily living even more.

Nevertheless, supervised individual tailored physical exercises, is a recommended non-pharmacological treatment of POTS. However, few studies have investigated the effect of physical exercise in POTS, and studies of POTS and post COVID-19 condition are very sparse. Therefore a feasibility study were performed and data found that the intervention (individually tailored physical exercise) was feasible in terms of safety, recruitment and compliance. Moreover the feasibility study provided optimistic results of the effects according to the participants physical, psychological functions as to their quality of life.

The planned RCT is part of research project (ReCOV), integrated with the clinical follow-up at Karolinska University Hospital and linked research project of patients who have been hospitalized or refereed to the clinic from primary care. The hypothesis is that an individually tailored rehabilitation program will have a beneficial effect on the ability to spend time in an upright position, as well as on HRQoL, for individuals with POTS, post COVID-19 condition.

The overall aim of this study is to evaluate the effects of an individually tailored exercise and its impact on time spent in upright position and health-related quality of life (HRQoL), physical activity, physical and psychological function and work-ability in persons with POTS, post COVID-19 condition.

Methods

Participants:

A total of 60 adult patients (>18 years) with POTS (diagnosed by a cardiologist), post COVID-19 condition. Recruitment will take place at the outpatient clinic at Karolinska University Hospital or in the primary care in Region Stockholm. Exclusion criteria: known pregnancy, cancer, already ongoing individual physical exercise (specific for POTS) or not able to perform measurements and/or intervention.

Procedure:

Prior to randomization baseline measurements will be performed. The measurements include Active Standing (AST), Test, 6-minute Walk Test (6MWT), muscle strength with MicroFET, measurements of pulsoximetry, pulse and blood pressure before, during and after tests, and participant will report their symptoms with BORG CR10 and BORG RPE. To evaluate time in upright position participants will wear two accelerometers (ActivPAL) during a week before intervention start. Questionnaires that will be used are EQ-5D-5L, Vanderbuildt Orthostatic Symptom Scale (VOSS), Malmö POTS Symptom Scale (MaPS), Fatigue Severeity Scale (FSS), Mental Fatigue Scale (MFS), DePaul Symtom Questionnaire - Post-Exertion Malaise (DSQ-PEM), Generalized Anxiety Disorder 7-item scale (GAD-7), Patient Health Questionnaire (PHQ-9) and Insomnia Severeity Index (ISS).

Controls: Participants randomized to control will receive standard care during 16 weeks. Standard care includes (but not restricted to) information about POTS and lifestyle changes that may effect the symptoms, advice about what fluid intake and nutrition, compression garments, pharmacological interventions etc.

Intervention: Participants randomized to intervention will receive standard care (same as controls) and undergo an individually tailored physical exercise program during a period of 16 weeks. The intervention will consist of exercises to enhance muscle strength and endurance. The program includes progression regarding duration and position for the exercise (starting i laying position and progression towards upright position). Progression should be halted if post exertional malaise (PEM) or other problems occur whitin 24h after exercise. The participants will once a week be supervised and guided individually by a physioherapist. Participants will, on a weekly basis, complete a training diary regarding their physical activity and training intensity in which they report any setbacks or adverse events.

Measurements of both groups (control and intervention) will be repeated after completion of a period of 16 weeks and longitudinal follow-up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) diagnosed with POTS (by a cardiologist) post COVID-19 condition.

Exclusion Criteria:

* known pregnancy, cancer, already ongoing intervention of individual tailored physical exercise as the intervention (specific for POTS), unable to perform measurements and/or intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in time in upright position and steps per day | through study completion, an average of 1 year
  Measured with two accelerometers, one attached to the chest and one to the lower limbs, to measure time (hours, minutes) in upright position
Change in Health-Related Quality of Life (HRQoL) | through study completion, an average of 1 year
  Measured with EuroQualityOf Life 5 dimensions questionnaire (EQ-5D-5L), which is an instrument that evaluates the generic quality of life. EQ-5D includes a descriptive system, which comprises 5 dimensions of health: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. A descriptive index-score between 0-1, higher score indicates higher HRQoL. EQ-5D also includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher HRQoL.

SECONDARY OUTCOMES:
Change in walking distance during 6 minute walk test | through study completion, an average of 1 year
  Change in walking distance measured in meters during 6 minutes walk test (6MWT)
Change in oxygen saturation during 6 minute walk test | through study completion, an average of 1 year
  Change in the lowest oxygen saturation level measured in percentage (%) with pulse oximetry during 6 minute walk test
Change in dyspnea during 6 minute walk test | through study completion, an average of 1 year
  Change in perceived dyspnea measured with Borg Category-Ratio scale (Borg CR-10) at the end of 6 minute walk test. Borg CR-10 ranging between 0-10. The higher the score, the higher the dyspnea.
  calculated by subtracting the oxygen level at rest before the test with the lowest level during the test.
Change in leg fatigue during 6 minute walk test | through study completion, an average of 1 year
  Change in perceived leg fatigue measured with Borg CR-10 at the end of 6 minute walk test. Borg CR-10 ranging between 0-10. The higher the score, the higher the leg fatigue. test. Borg CR-10 ranging between 0-10. The higher the score, the higher the dyspnea.
  calculated by subtracting the oxygen level at rest before the test with the lowest level during the test.
Change in exertion during 6 minute walk test | through study completion, an average of 1 year
  Change in perceived exertion measured with Borg Rating of Perceived Exertion (Borg RPE) at the end of 6 minutes walk test. Borg RPE ranging between 6-20. The higher the score, the higher the exertion.
Change in heart rate during 6 minute walk test | through study completion, an average of 1 year
  Change in the highest heart rate measured in beats per minute with pulseoxymeter during 6 minute walk test
Change in Self-reported POTS-symptoms | through study completion, an average of 1 year
  Measured with Malmö-POTS-questionnaire (MaPS), which is a self assessment tool examining common symptoms in POTS. MaPS consists of 12 items. Patients are asked to rate symptoms on a scale from 0-10 on each item. 0 i= no symptom and 10 = worst imaginable. Total score ranging from 0-120. Higher score indicates more POTS-symptoms.
Change in Anxiety - Generalised Anxiety Disorder 7-item scale | through study completion, an average of 1 year
  Measured with Generalised Anxiety Disorder 7-item scale (GAD-7) which is a self assessment tool. Total score ranging from 0-21. Higher score indicates higher anxiety.
Change in Depression - Patient Health Questionnaire-9 | through study completion, an average of 1 year
  Measured with Patient Health Questionnaire-9 (PHQ-9). PHQ-9 which contains 9 items. Total score ranges from 0 to 27. Higher score indicate more severe depression symptoms
Change in Fatigue | through study completion, an average of 1 year
  Measured with Fatigue Severity Scale (FSS), which is a 9-item scale that measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Total score ranging from 9-63. The higher the score, the more severe the fatigue is. Fatigue also measured with Mental Fatigue Scale (MFS), which is a 15-item scale that measures the severity of mental fatigue. Total score ranging from 0-44. The higher the score, the more severe the fatigue is.
Change in Self-reported outcome measure of physical function | through study completion, an average of 1 year
  Measured with Patient Specific Functional Scale (PSFS), a questionnaire that can be used to quantify activity limitation and measure functional outcome for patients. Patients are asked to identify three to five important activities they are unable to perform or are having difficulty with because of their problem. In addition to identifying the activities, patients are asked to rate, on a scale ranging from 0-10, the current level of difficulty associated with each activity. The higher the score, the less difficulty to perform the activity
Change in blood pressure during Active standing test | through study completion, an average of 1 year
  Measured with Active standing test according to a specific protocol with measurements of responses in systolic and diastolic blood pressure after getting up to standing from the supine position
Change in heart rate response during Active standing test | through study completion, an average of 1 year
  Measured with Active standing test according to a specific protocol with measurements of responses in heart rate after getting up to standing from the supine position.
Change in oxygen saturation during Active standing test | through study completion, an average of 1 year
  Measured with Active standing test according to a specific protocol with measurements of responses in oxygen saturation, measured with pulse oximetry, after getting up to standing from the supine position.
Change in respiratory rate during Active Standing Test | through study completion, an average of 1 year
  Change in respiratory rate, measured in number of breaths/min before and after the Active Standing Test
Change in dyspnea during Active standing test | through study completion, an average of 1 year
  Measured with Active standing test according to a specific protocol with measurements of responses in perceived dyspnea measured with Borg CR-10 scale after getting up to standing from the supine position.
Change in leg fatigue during Active Standing Test | through study completion, an average of 1 year
  Change in perceived leg fatigue measured with Borg CR-10 before, during and at the end of Active Standing Test.
Change in exertion during Active standing test | through study completion, an average of 1 year
  Measured with Active standing test according to a specific protocol with measurements of responses in perceived exertion with Borg RPE scale after getting up to standing from the supine position.
Change in Physical activity | through study completion, an average of 1 year
  Measured with Frändin/Grimby activity scale, which is a self-assessment scale about current levels of physical activity, ranging from 1 to 6. The higher the score, the higher the level of physical activity
Change in orthostatic symptoms | through study completion, an average of 1 year
  Assessed with the Vanderbilt Orthostatic Symptom Scale (VOSS). After the Active standing test (AST) the participant uses a self-assessment questionnaire about orthostatic symptoms prominent during the Active standing test (performed according to a specific protocol with measurements of responses in systolic and diastolic blood pressure after getting up to standing from the supine position). The scale range from 0=no symptoms, to 10=worst imaginable symptoms. The scale includes 9 items regarding orthostatic symptoms and the higher the score, the higher level of symptoms during the orthostatic test.
Change in insomnia | through study completion, an average of 1 year
  Measured with Insomnia Severity Index (ISI), a 7-item questionnaire. Score between 0-28, with higher score indication a more severe insomnia.
Change in Workability | through study completion, an average of 1 year
  Measured in percentage of full time work, ranging from 0-100%
Change in muscle strength | through study completion, an average of 1 year
  Measured with the wireless microFET®2 Digital Handheld Dynamometer muscle tester. measurements of isometric muscle strength will be carried out on muscles in the lower extremity according to guidelines.
Change in post-exertional-Malaise (PEM) | through study completion, an average of 1 year
  Measured by the quiestionnaire; DePaul Symptom Questionnaire-Post Exertional Malaise Short-form (DSQ-PEM). DSQ-PEM is a 10 item questionnaire that includes scoring of frequency and severity of PEM and indicate if ME/CFS may be present. Higher score indicates more severe PEM.
Change in pharmacological treatment of POTS | through study completion, an average of 1 year
  Assessed by gathering information from the participants and from their medical journal of what type of pharmacological treatment they're in need of and the dose.
Compliance to intervention | through study completion, an average of 1 year
  Assessed by participant diaries during 16weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malin Nygren-Bonnier, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu Q, Levine BD. Exercise and non-pharmacological treatment of POTS. Auton Neurosci. 2018 Dec;215:20-27. doi: 10.1016/j.autneu.2018.07.001. Epub 2018 Jul 4. PMID 30001836
- [Background] Crook H, Raza S, Nowell J, Young M, Edison P. Long covid-mechanisms, risk factors, and management. BMJ. 2021 Jul 26;374:n1648. doi: 10.1136/bmj.n1648. PMID 34312178
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Fedorowski A. Postural orthostatic tachycardia syndrome: clinical presentation, aetiology and management. J Intern Med. 2019 Apr;285(4):352-366. doi: 10.1111/joim.12852. Epub 2018 Nov 23. PMID 30372565
- [Background] Johansson M, Stahlberg M, Runold M, Nygren-Bonnier M, Nilsson J, Olshansky B, Bruchfeld J, Fedorowski A. Long-Haul Post-COVID-19 Symptoms Presenting as a Variant of Postural Orthostatic Tachycardia Syndrome: The Swedish Experience. JACC Case Rep. 2021 Apr;3(4):573-580. doi: 10.1016/j.jaccas.2021.01.009. Epub 2021 Mar 10. PMID 33723532
- [Background] Stahlberg M, Reistam U, Fedorowski A, Villacorta H, Horiuchi Y, Bax J, Pitt B, Matskeplishvili S, Luscher TF, Weichert I, Thani KB, Maisel A. Post-COVID-19 Tachycardia Syndrome: A Distinct Phenotype of Post-Acute COVID-19 Syndrome. Am J Med. 2021 Dec;134(12):1451-1456. doi: 10.1016/j.amjmed.2021.07.004. Epub 2021 Aug 11. PMID 34390682
- [Background] Arnold AC, Ng J, Raj SR. Postural tachycardia syndrome - Diagnosis, physiology, and prognosis. Auton Neurosci. 2018 Dec;215:3-11. doi: 10.1016/j.autneu.2018.02.005. Epub 2018 Feb 28. PMID 29523389
- [Background] Benrud-Larson LM, Dewar MS, Sandroni P, Rummans TA, Haythornthwaite JA, Low PA. Quality of life in patients with postural tachycardia syndrome. Mayo Clin Proc. 2002 Jun;77(6):531-7. doi: 10.4065/77.6.531. PMID 12059122